CLINICAL TRIAL: NCT05774405
Title: Short-term Effects of Transdermal Estradiol on Female COVID-19 Patients: A Randomized Placebo-Controlled Study
Brief Title: Short-term Effects of Transdermal Estradiol on Female COVID-19 Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Turkish Menopause and Osteoporosis Society (Unknown); Karakoy Rotary Club (Unknown); Rebul Pharmacy (Unknown)
Responsible Party: Principal Investigator, Cemal Tamer Erel, Clinical Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 68871907-604.01.01-67414
Record Dates: First submitted 2023-03-15; First posted 2023-03-17 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; Hormone Replacement Therapy
Keywords: Covid-19; hormone replacement therapy
MeSH Terms: conditions — COVID-19 | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): All patients were treated with favipiravir for a week. At the same time, the patients in this arm received Estradiol patch (Climara 7.8 mg patch/week, Bayer, Germany) for 14 days.
  Interventions: Drug: Climara 0.1Mg/24Hr Transdermal System
- Placebo (Placebo Comparator): All patients were treated with favipiravir for a week. At the same time, the patients in this arm received Hydrogel patch (Adhesive Hydrogel patch/week, Rebul Pharmacy, Turkey) for 14 days.
  Interventions: Other: Hydrogel patch

INTERVENTIONS:
Drug: Climara 0.1Mg/24Hr Transdermal System — Transdermal estradiol patch is used.
  Arms: Experimental
Other: Hydrogel patch — Adhesive Hydrogel patch
  Arms: Placebo

SUMMARY:
The goal of this randomized placebo-controlled study is to investigate the short-term effects of transdermal estrogen therapy on postmenopausal women with COVID-19 disease.

The main question[s] it aims to answer are:

* the clinical outcomes with adding estrogen treatment to conventional therapy of Covid-19 disease
* the biochemical outcomes with adding estrogen treatment to conventional therapy of Covid-19 disease

All participants received favipiravir for a week according to the national guidelines published by the Health Ministry of Turkish Republic at that time.

As an intervention, transdermal estradiol patch (7.8 mg patch/week) was applied for 14 days on the upper buttock of the patients in experimental arm. As a placebo, hydrogel patch (adhesive hydrogel patch/week) was applied to the female patients for 14 days.

Researchers compared experimental and control groups to see if the impact of adding estrogen on the clinical course of Covid-19 disease

DETAILED DESCRIPTION:
The risk of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, morbidity and mortality from Covid-19 disease were higher among men compared to women. This is caused by the differences in immunological response and viral pathogenesis between men and women. It is theoretically assumed that estrogen has a positive impact on female COVID-19 patients. In this randomized placebo-controlled study, we aimed to investigate the short-term effects of transdermal estrogen therapy on postmenopausal women with COVID-19 disease. Female patients diagnosed with Covid-19 disease were examined and only postmenopausal women were included into the study. The COVID-19 diagnosis was made with a positive reverse transcription-polymerase chain reaction (RT-PCR) test given with nasal and oral swabs. All participants received favipiravir for a week according to the national guidelines published by the Health Ministry of Turkish Republic at that time.

As an intervention, transdermal estradiol patch (7.8 mg patch/week) was applied for 14 days on the upper buttock of the patients in experimental arm. As a placebo, hydrogel patch (adhesive hydrogel patch/week) was applied to the female patients for 14 days.

Our primary outcome was to achieve better clinical and biochemical outcomes with adding estrogen treatment to conventional therapy of Covid-19 disease. The epidemiological and clinical data, the results of biochemical analysis, the information regarding the treatment and outcomes and serum estradiol levels were determined.

ELIGIBILITY:
Inclusion Criteria:

* Female patients diagnosed with Covid-19 disease
* Postmenopausal women (who had 12 months of amenorrhea after their final menstrual period)
* Positive reverse transcription-polymerase chain reaction (RT-PCR) test given with nasal and oral swabs

Exclusion Criteria:

* Negative RT-PCR test
* Female patients at reproductive stage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9169 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Evidence of disease progression for mild cases | 15 days
  Proportion of patients who are hospitalised in 15 days
Evidence of disease progression for moderate and severe cases | 15 days
  Proportion of patients who required mechanical ventilation or died within 15 days
Kidney function tests | 15 days
  change of urea(mg/dL), creatinine(mg/dL) and uric acid (mg/dL) levels with estrogen and hydrogel patch application
Platelet | 15 days
  change of platelets in total blood count (*10^3/μL) with estrogen and hydrogel patch application
Markers of coagulation | 15 days
  change of fibrinogen (mg/dL) and D-dimer (mg/L) with estrogen and hydrogel patch application
Marker of inflammation | 15 days
  change of C-reactive protein (mg/L) levels within 15 days

SECONDARY OUTCOMES:
serum E2 levels | 15 days
  change of serum E2 levels with estrogen and hydrogel patch application
rate of death | 15 days
  comparison of rate of death in each arm
rate of complications | 15 days
  comparison of rate of complications in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Cemal Tamer Erel, Prof, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No